CLINICAL TRIAL: NCT04141930
Title: Pilot of Cohort of Households for Influenza Monitoring and Evaluation in Seattle (pCHIMES)
Brief Title: Pilot of Cohort of Households for Influenza Monitoring and Evaluation in Seattle
Acronym: pCHIMES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Helen Chu, Assistant Professor, School of Medicine: Allergy and Infectious Diseases, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008200
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Influenza; Respiratory Viral Infection
Keywords: influenza; flu; antiviral; baloxavir; Xofluza; rapid delivery; self-test
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Drug Eligible (Other): Baloxavir given in 40 mg and 80 mg tablets for single-dose oral consumption during the first influenza infection for that participant
  Interventions: Drug: Baloxavir Marboxil

INTERVENTIONS:
Drug: Baloxavir Marboxil — Individuals willing and able, will receive a weight-based oral dose of baloxavir within 48 hours of symptom onset
  Other Names: Xofluza

SUMMARY:
This study will evaluate a home-based approach to influenza infection control, using prepositioned home-based influenza self-test kits, telemedicine services, and rapid delivery of Xofluza (Baloxavir marboxil) for administration within 48 hours of symptom onset.

DETAILED DESCRIPTION:
Households represent an important location for transmission of influenza. Rapid delivery of Xofluza may reduce household exposures to influenza among susceptible individuals.This study is a pilot study of a home-based approach to influenza infection control, utilizing self-test kits and rapid home delivery of an antiviral. Households with at least 3 individuals residing there at least 4 days a week, including at least 2 household members that are eligible to take antiviral, will be monitored throughout the influenza season for the onset of a cough or two or more acute respiratory infection symptoms. This study will be conducted in households in the Seattle, WA area for one influenza season, beginning November 1, 2019 and ending April 1, 2020. Household will self-monitor for onset of symptoms throughout the influenza season. When symptoms develop, the participant will self-test for influenza infection using a prepositioned home-testing kit. If negative, the ill participant will provide one self-collected nasal swab specimen. If positive, the ill participant will connect with a healthcare provider via the tele-health app on their smartphone to confirm the influenza diagnosis. Next, if eligible to receive Xofluza, the influenza-positive individual will receive a rapid home delivery of Xofluza within 2-6 hours of the positive test result. All influenza-positive participants will provide a self-collected nasal swab specimen at Study Day 0, Study Day 2-3, and Study Day 5-7. For all illness episodes, the ill individual will complete a questionnaire regarding symptom duration and severity, as well as behavioral changes due to illness.

ELIGIBILITY:
Inclusion Criteria:

* Household Level:
* Group of at least 3 individuals of any ages defined as at least 3 persons residing at the same address for at least 4 days per calendar week
* Household group utilizes common household areas
* At least 2 household members meeting all individual inclusion/exclusion criteria listed below and willing to participate (e.g. at least two members of the household are 12 years of age or older)
* At least one member of the household has a smartphone
* Individual Level: Drug Eligible
* Resident of a household with 3 or more members (including eligible cases) for 4 or more days a calendar week
* Age 12 years or older weighing at least 40 kg (greater than 88 pounds)
* Willing and able to take study medication
* Willing to comply with all study procedures
* English-speaking
* Able to provide written, informed consent and/or assent (if applicable)
* Permanent mailing address that is available for study staff to mail necessary materials
* Individual Level: Drug Ineligible
* Resident of a household with 3 or more members (including eligible cases) for 4 or more days a calendar week
* Willing to comply with all study procedures
* English-speaking
* Able to provide written, informed consent and/or assent (if applicable)

Exclusion Criteria:

* Household Level:
* Previous documentation of an influenza infection prior to or during the annual influenza season in any household member prior to enrollment
* Individual Level:
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration
* Individuals with hypersensitivity to baloxavir
* Individuals that already have a tele-health account
* Any individual that has one or more of the following conditions:
* Pregnant
* Currently lactating
* Immunosuppressed or immunocompromised (by disease or medication)
* Cancer
* Liver disease
* Kidney disease

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Y Chu, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We do not currently expect to share specimens with outside investigators, but if compelling opportunities arise that will advance the overall objectives of this research, the Executive Committee of the study will consider such requests. They alone have the authority to make such decisions.
  All biospecimens (nasal swabs) will be coded and identifiable through the study's main database. Any specimens shared with external investigators (if deemed appropriate by the Executive Committee) will have identifiers removed prior to sharing.

REFERENCES:
- [Background] Hayden FG, Sugaya N, Hirotsu N, Lee N, de Jong MD, Hurt AC, Ishida T, Sekino H, Yamada K, Portsmouth S, Kawaguchi K, Shishido T, Arai M, Tsuchiya K, Uehara T, Watanabe A; Baloxavir Marboxil Investigators Group. Baloxavir Marboxil for Uncomplicated Influenza in Adults and Adolescents. N Engl J Med. 2018 Sep 6;379(10):913-923. doi: 10.1056/NEJMoa1716197. PMID 30184455
- [Background] Hayden FG, Belshe R, Villanueva C, Lanno R, Hughes C, Small I, Dutkowski R, Ward P, Carr J. Management of influenza in households: a prospective, randomized comparison of oseltamivir treatment with or without postexposure prophylaxis. J Infect Dis. 2004 Feb 1;189(3):440-9. doi: 10.1086/381128. Epub 2004 Jan 26. PMID 14745701
- [Background] Welliver R, Monto AS, Carewicz O, Schatteman E, Hassman M, Hedrick J, Jackson HC, Huson L, Ward P, Oxford JS; Oseltamivir Post Exposure Prophylaxis Investigator Group. Effectiveness of oseltamivir in preventing influenza in household contacts: a randomized controlled trial. JAMA. 2001 Feb 14;285(6):748-54. doi: 10.1001/jama.285.6.748. PMID 11176912
- [Background] Leung YH, Li MP, Chuang SK. A school outbreak of pandemic (H1N1) 2009 infection: assessment of secondary household transmission and the protective role of oseltamivir. Epidemiol Infect. 2011 Jan;139(1):41-4. doi: 10.1017/S0950268810001445. Epub 2010 Jun 21. PMID 20561390
- [Background] Fry AM, Goswami D, Nahar K, Sharmin AT, Rahman M, Gubareva L, Azim T, Bresee J, Luby SP, Brooks WA. Efficacy of oseltamivir treatment started within 5 days of symptom onset to reduce influenza illness duration and virus shedding in an urban setting in Bangladesh: a randomised placebo-controlled trial. Lancet Infect Dis. 2014 Feb;14(2):109-18. doi: 10.1016/S1473-3099(13)70267-6. Epub 2013 Nov 22. PMID 24268590
- [Background] Takashita E, Ichikawa M, Morita H, Ogawa R, Fujisaki S, Shirakura M, Miura H, Nakamura K, Kishida N, Kuwahara T, Sugawara H, Sato A, Akimoto M, Mitamura K, Abe T, Yamazaki M, Watanabe S, Hasegawa H, Odagiri T. Human-to-Human Transmission of Influenza A(H3N2) Virus with Reduced Susceptibility to Baloxavir, Japan, February 2019. Emerg Infect Dis. 2019 Nov;25(11):2108-2111. doi: 10.3201/eid2511.190757. Epub 2019 Nov 17. PMID 31436527
- [Derived] Emanuels A, Casto AM, Heimonen J, O'Hanlon J, Chow EJ, Ogokeh C, Rolfes MA, Han PD, Hughes JP, Uyeki TM, Frazar C, Chung E, Starita LM, Englund JA, Chu HY; Seattle Flu Study Investigators. Remote surveillance and detection of SARS-CoV-2 transmission among household members in King County, Washington. BMC Infect Dis. 2024 Mar 13;24(1):309. doi: 10.1186/s12879-024-09160-z. PMID 38481147

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug Eligible: Baloxavir given in 40 mg and 80 mg tablets for single-dose oral consumption during the first influenza infection for that participant. Individuals need to be eligible based on on-label use according to their age and medical history.
  Baloxavir Marboxil: Individuals willing and able, will receive a weight-based oral dose of baloxavir within 48 hours of symptom onset
- Study Drug Ineligible: Individuals not eligible to receive on-label use of Baloxavir due to age or medical history
Period: Overall Study
Arm/Group | Study Drug Eligible | Study Drug Ineligible
Started | 302 | 179 (The 179 individuals that were not eligible to receive the study drug, participated in an observation portion of the study where all study procedures were the same excluding telehealth visit and an antiviral delivery.)
Completed | 302 | 179
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on individuals that contributed data during the test-and-treat phase of the protocol.
Arm/Group | Study Drug Eligible
Number analyzed (Participants) | 481
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 221
  Between 18 and 65 years | 250
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253
  Male | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35
  Not Hispanic or Latino | 439
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 408
  More than one race | 31
  Unknown or Not Reported | 23
Region of Enrollment [Number; unit: participants]
  United States | 481

OUTCOME MEASURES:

1. Primary Outcome: Initiate Antiviral Therapy Within 48 Hours of Symptom Onset
Description: Among symptomatic participants, this outcome measure will be calculated by determining the number of home influenza test-positive, drug eligible participants that were prescribed and rapidly delivered baloxavir by the study within 48 hours of symptom onset.
Time Frame: Up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug Eligible
Number analyzed (Participants) | 8
Participants | 8

2. Secondary Outcome: Home Influenza Tests Confirmed by Laboratory Testing
Description: Proportion of individuals who test positive for influenza using the home-based influenza test compared to the number of individuals that test positive for influenza via a PCR laboratory test
Time Frame: Up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug Eligible
Number analyzed (Participants) | 12
Participants | 8

3. Secondary Outcome: Delivered Antivirals Within 48 Hours of Symptom Onset
Description: Proportion of individuals who are delivered antivirals within 48 hours of symptom onset. Only drug eligible study participants prescribed an antiviral
Time Frame: Up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug Eligible
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 14 days after receipt of antiviral
Arm/Group | Study Drug Eligible
All-Cause Mortality (participants affected / at risk) | 0/302
Serious Adverse Events (participants affected / at risk) | 1/302
Other Adverse Events (participants affected / at risk) | 5/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug Eligible (N=302)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug Eligible (N=302)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Headache (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04141930/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04141930/SAP_001.pdf